CLINICAL TRIAL: NCT02938611
Title: Feasibility Study on Estimating the Prevalence and Management of Stage 4 Chronic Kidney Disease in Adults Via Laboratories and Nephrologists in the Gard, France
Brief Title: Feasibility of Estimating the Prevalence and Management of Stage 4 CKD the Gard, France
Acronym: MRC-Gard
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2016-06/OM-01
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: Persons with stage >=4 chronic kidney disease.

SUMMARY:
The main objective of this study is to evaluate the feasibility of estimating the prevalence of stage 4 and 5 chronic kidney disease in the Gard department of France from data obtained via laboratory databases. To verifiy if the demand for care thus authenticated by laboratory tests is adapted to nephrology care delivery, as recommended by the French High Authority of Health (HAS), laboratory data will be compared with those of patients seen by nephrologists in the department.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease (stage >= 4)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with >= stage 4 chronic kidney disease and residing in the Gard department of France.
Sampling Method: Probability Sample
Enrollment: 3375 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of chronic kidney disease stage > = 4 in the Gard according to laboratory data (raw number) | from baseline (day 0) to 12 months
The prevalence of chronic kidney disease stage > = 4 in the Gard according to laboratory data (%) | from baseline (day 0) to 12 months

SECONDARY OUTCOMES:
The percentage of patients with CKD stage >= 4 correctly reported by participating nephrologists | from baseline (day 0) to 12 months
For each nephrologist participating in the study, the % of patients with stage >=4 chronic kidney disease who are correctly declared | from baseline (day 0) to 12 months
The % of patients with chronic kidney disease stage > = 4 in the Gard according to laboratory data and who are not seen by a nephrologist | from baseline (day 0) to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moranne, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - AIDER - Unité de Dialyse d'Alès, Alès
  - AIDER - Unité de Dialyse de Nîmes, CHU Carémeau, Nîmes
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Gardialyse, Nîmes